CLINICAL TRIAL: NCT05216094
Title: Effects of Applying Task-oriented Practice Combined With Behavior Changes Strategy and Mhealth App on the Improvement of Upper Limb Function for Patients With Chronic Stroke
Brief Title: Effects of Mhealth App on the Improvement of Upper Limb Function for Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-E(I)-20200437
Record Dates: First submitted 2022-01-24; First posted 2022-01-31 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2022-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smart phone intervention group (Experimental): smart phone intervention group stroke subjects completed smart phone App tasks with affected upper limb or bilateral arm movement for 12 weeks
  Interventions: Other: smart phone App
- conventional group (Active Comparator): stroke subjects receive conventional rehabilitation home program for 12 weeks
  Interventions: Other: conventional rehabilitation

INTERVENTIONS:
Other: smart phone App — stroke subjects completed tasks-oriented program demoed in the smart phone app with affected upper limb or bilateral arm movement for 12 weeks
  Arms: smart phone intervention group
Other: conventional rehabilitation — stroke subjects receive conventional rehabilitation home program with smart phone app ,without task-oriented program demoed function, for 12 weeks
  Arms: conventional group

SUMMARY:
The main purpose is to develop a mobile health app that combines behavioral change technology and task-oriented exercise strategies to provide a technology-assisted training system for upper limb motor function in home stroke cases, and to analyze its feasibility and therapeutic benefits. It is estimated that 50 chronic stroke cases will be recruited and randomly assigned to the experimental group (n=25) and the control group (n=25). The experimental group received a 12-week action health App combined with behavioral change technology and task-oriented upper limb exercise strategy intervention. The control group received a 12-week sham control and a traditional home rehabilitation intervention program. Both groups received pre-test, post-test (12 weeks) and follow-up assessment (4 weeks). This study will adopt a double-blind evaluation design.

DETAILED DESCRIPTION:
The main purpose is to develop a mobile health app that combines behavioral change technology and task-oriented exercise strategies to provide a technology-assisted training system for upper limb motor function in home stroke cases, and to analyze its feasibility and therapeutic benefits. It is estimated that 50 chronic stroke cases will be recruited and randomly assigned to the experimental group (n=25) and the control group (n=25). The experimental group received a 12-week action health App combined with behavioral change technology and task-oriented upper limb exercise strategy intervention. The control group received a 12-week sham control and a traditional home rehabilitation intervention program. Both groups received pre-test, post-test (12 weeks) and follow-up assessment (4 weeks). This study will adopt a double-blind evaluation design, and the evaluation contents include Fugl-Meyer Upper Limb Motor Function Scale, Grip Strength Assessment, Box and Block Test, MAL-28, Stroke Impact Scale and System Utility Scale. Data analysis included descriptive statistics, Repeated ANOVA, and correlation analysis.

The results of this research are expected to develop a mobile health app that combines behavioral change technology and task-oriented exercise strategies, which can be applied to stroke patients at home or in the community to promote the execution of high-intensity and high-repetition upper limb motor function exercises, thereby improving upper limb and daily life. life function.

ELIGIBILITY:
Inclusion Criteria:

* Age >20, and first onset
* Unilateral Hemiplegia
* No obvious cognitive impairment (Mini-Mental State Examination (MMSE) score > 23)
* The FMA upper limb movement score is above 30 points, and there are partial extension movements of the affected fingers and wrists
* Ability to operate a smartphone independently before or at present
* Those who have no obvious vision loss and can read mobile phone text clearly

Exclusion Criteria:

* Language barriers or aphasia
* Other orthopedic diseases (such as severe shoulder pain, joint contractures) or nerve damage (such as peripheral nerve damage) that affect the movement of the upper limbs
* People with abnormal cardiopulmonary function who are not suitable for active sports
* Feel severe Absence, FMA sensory score <12 points
* Other progressive diseases such as cancer, amyotrophic lateral sclerosis, multiple sclerosis, etc

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Box and Block Test | pre-test, post-test(Change from pre-test Box and Block Test after 12 weeks' intervention), and follow-up(Change from post-test Box and Block Test at one month )
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke.
FUGL-MEYER ASSESSMENT-UE, FMA) | pre-test, post-test(Change from pre-test FUGL-MEYER ASSESSMENT-UE after 12 weeks' intervention), and follow-up(Change from post-test FUGL-MEYER ASSESSMENT-UE at one month )
  Fugl-Meyer Assessment (FMA) scale is an index to assess the sensorimotor impairment in individuals who have had stroke.
Grip Strength Assessment | pre-test, post-test(Change from pre-test Grip Strength Assessment after 12 weeks' intervention), and follow-up(Change from post-test Grip Strength Assessment at one month )
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength.
System Usability Scale(SUS) | only post-test(after 12 weeks' intervention)
  The System Usability Scale, is a simple survey that provides a high-level score for the usability of a product. The score is a value between 0 and 100, with higher values indicating better usability.
Motor Activity Log (MAL-28) | pre-test, post-test(Change from pre-test Motor Activity Log after 12 weeks' intervention), and follow-up(Change from post-test Motor Activity Log at one month )
  The Motor Activity Log (MAL) is a subjective measure of an individual's real life functional upper limb performance.
Stroke Impact Scale(SIS) | pre-test, post-test(Change from pre-test Stroke Impact Scale after 12 weeks' intervention), and follow-up(Change from post-test Stroke Impact Scale at one month )
  The purpose of this questionnaire is to evaluate how stroke has impacted your health and life. The score is a value between 0 and 100, with higher values indicating better recover.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Jong Chang, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Department of Occupational Therapy, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: starting one year after publication
Access Criteria: For Meta-analysis study

REFERENCES:
- [Result] Szturm T, Imran Z, Pooyania S, Kanitkar A, Mahana B. Evaluation of a Game Based Tele Rehabilitation Platform for In-Home Therapy of Hand-Arm Function Post Stroke: Feasibility Study. PM R. 2021 Jan;13(1):45-54. doi: 10.1002/pmrj.12354. Epub 2020 Apr 13. PMID 32107868
- See also: Evaluation of a Game Based Tele Rehabilitation Platform for In-Home Therapy of Hand-Arm Function Post Stroke: Feasibility Study — https://pubmed.ncbi.nlm.nih.gov/32107868/